CLINICAL TRIAL: NCT07167914
Title: A Phase 1 Study to Assess Safety, Tolerability and Pharmacokinetics of Single and Multiple Transdermal Doses of SFG-02 in Japanese and White Healthy Adult Participants
Brief Title: A Study to Assess Safety, Tolerability and Pharmacokinetics of Transdermal SFG-02 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juro Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SFG-02-101
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Health Participants
Keywords: White Healthy Participants; Japanese Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- (1) SFG-02 Single Transdermal Application (Experimental): Assign 8 Japanese Participants for SFG-02 or Placebo Application
  Interventions: Drug: SFG-02; Drug: Placebo
- (2) SFG-02 (1st) Repeated Transdermal Application for 10 days (Experimental): Assign 8 Japanese Participants for SFG-02 1st Dose or Placebo Application (10 days)
  Interventions: Drug: SFG-02; Drug: Placebo
- (3) SFG-02 (2nd) Repeated Transdermal Application for 10 days (Experimental): Assign 8 Japanese Participants for SFG-02 2nd Dose or Placebo Application (10 days)
  Interventions: Drug: SFG-02; Drug: Placebo
- (4) SFG-02 Single Transdermal Application (White) (Experimental): Assign 8 White Participants for SFG-02 or Placebo Application (single)
  Interventions: Drug: SFG-02; Drug: Placebo

INTERVENTIONS:
Drug: SFG-02 — Transdermal Formulation (SFG-02)
Drug: Placebo — Transdermal Formulation (Placebo)

SUMMARY:
This Phase 1 study will evaluate the safety, tolerability, and pharmacokinetics of a novel transdermal formulation of SFG-02 following single and repeated applications in Japanese and White healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese or white male and female participants aged between 18 and 45 years at the time of consent.
2. Participants who agree to use contraception during a specified period.
3. Participants with a Body Mass Index (BMI) of at least 18.0 kg/m2 and less than 32.0 kg/m2.
4. Participants who are judged to be healthy by the principal (or sub-) investigator.
5. Participants must understand the methods and compliance requirements of this study and must give his/her free and voluntary written consent to participate in this study.

Exclusion Criteria:

1. Participants with clinically relevant symptoms, diseases, or pre-existing conditions.
2. Participants with extensive skin findings on the abdomen.
3. Participant who has used or will use prescription drugs, non-prescription drugs or products containing herbal medicines within a specified period
4. Participants whose normal weekly alcohol intake exceeds 150 g.
5. Habitual consumers of caffeine-containing beverages who are likely to experience symptoms if they stop.
6. Smokers or those who have smoked or used other nicotine-containing products within 6 months.
7. Participants who participated in a clinical trial and took a new active pharmacological ingredient within a specified period.
8. Participants who have undergone surgery within 4 weeks.
9. Pregnant or lactating women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | From the first application to the 14th day after the final application
  Incidence of Treatment-Emergent Adverse Events in Healthy Adult Subjects
Pharmacokinetics (PK): Maximum concentration (Cmax) of SFG-02 | At designated timepoints (up to 7 days after the final application)
  Blood samples will be collected at multiple timepoints to estimate Cmax of SFG-02
PK: Area under the concentration versus time curve (AUC) of SFG-02 | At designated timepoints (up to 7 days after the final application)
  Blood samples will be collected at multiple timepoints to estimate Tmax of SFG-02
PK: Time to maximum concentration (Tmax) of SFG-02 | At designated timepoints (up to 7 days after the final application)
  Blood samples will be collected at multiple timepoints to estimate Tmax of SFG-02
PK: Time to decrease the concentration by half (T1/2) of SFG-02 | At designated timepoints (up to 7 days after the final application)
  Blood samples will be collected at multiple timepoints to estimate T1/2 of SFG-02

CONTACTS AND LOCATIONS:
Locations (1):
- Sumida Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No